CLINICAL TRIAL: NCT02485977
Title: Cardiac MRI in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 15-16502
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary Hypertension: Adult patients with pulmonary hypertension referred for cardiac catheterization in the PI institution
  Interventions: Device: Magnetic resonance Imaging

INTERVENTIONS:
Device: Magnetic resonance Imaging — MRI study will be performed on 1.5 Tesla magnet, during the administration of Gadolinium

SUMMARY:
The overall goal of this study is to evaluate agreement between cardiac MR parameters and well-established clinical and catheterization parameters of poor prognosis in patients with pulmonary hypertension. The identification of noninvasive cardiac MR techniques to evaluate myocardial disease in patients with pulmonary hypertension would be beneficial to society due to the potential to replace serial invasive cardiac catheterization procedures with a noninvasive imaging test.

DETAILED DESCRIPTION:
1 BACKGROUND Currently the gold standard for evaluation of pulmonary hypertension is right heart pressure as measured by cardiac catheterization. Thus the method for stratifying patients with pulmonary hypertension in terms of risk and response to treatment is suboptimal, requiring multiple invasive procedures.

A number of studies have suggested that cardiac MR imaging is useful in the diagnosis of myocardial disease and may be related to patient prognosis in both ischemic and non-ischemic cardiomyopathy. Patients with pulmonary hypertension demonstrate post gadolinium delayed enhancement at the points of insertion of the right ventricle onto the inter-ventricular septum, and the presence of this finding has been shown to be inversely correlated with right ventricular function.

Quantitative evaluation of extracellular volume by post-gadolinium T1 relaxation time mapping (T1 mapping) and extracellular volume (ECV) mapping is used to quantify the extent of myocardial fibrosis, can detect fibrosis earlier than delayed enhancement imaging, and is particularly useful in non-ischemic or diffuse myocardial diseases. In addition, Displacement Encoding with Stimulated Echoes (DENSE) is a technique that allows quantification of tissue motion and myocardial strain, which can identify early myocardial dysfunction in patients with preserved ejection fraction, and therefore may be useful in the evaluation of myocardial function in pulmonary hypertension.

Utilization of novel cardiac MR techniques for quantitative assessment of the extent of subclinical myocardial disease in patients with pulmonary hypertension may therefore serve as a non-invasive tool to inform prognosis and surrogate biomarker to evaluate effectiveness of treatment strategies, with the potential to replace serial cardiac catheterization in these patients.

Our hypothesis is that utilization of novel cardiac MR techniques for quantitative assessment of the extent of subclinical myocardial disease in patients with pulmonary hypertension may serve as a non-invasive tool to inform prognosis and surrogate biomarker to evaluate effectiveness of treatment strategies, with the potential to replace serial cardiac catheterization in these patients.

Adult patients with pulmonary hypertension under clinical care at the UCSF pulmonary hypertension clinic who are referred for right heart catheterization will be invited to participate in our study. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Each participant will undergo cardiac MR examination during a single one-hour study visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Pulmonary hypertension

Exclusion Criteria:

* Pacemaker
* Renal dysfunction
* Cochlear implant
* Previous lung transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pulmonary hypertension referred for cardiac catheterization at UCSF
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
MRI scar burden measured by T1 mapping | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Medical Center, San Francisco, California, United States